CLINICAL TRIAL: NCT03210389
Title: A Prospective, Single-arm, and Open Clinical Trial of Chemotherapy With Lobaplatin and 5-FU on Efficacy and Safety in Recurrent Local or Distant Advanced NPC.
Brief Title: A Clinical Trial of Chemotherapy With Lobaplatin and 5-FU in Recurrent Local or Distant Advanced NPC.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yun-fei Xia, Director of Department of Radiation Oncology, Principal Investigator, Clinical Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2016-001-01
Record Dates: First submitted 2017-06-21; First posted 2017-07-06 (Actual); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Recurrent Nasopharyngeal Carcinoma
Keywords: Recurrent Nasopharyngeal Carcinoma; lobaptin
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — lobaplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- lobaplatin+5-FU (Experimental): Patients enrolled in this trial would get 4-6 cycles of lobaplatin + 5-FU chemotherapy.
  Interventions: Drug: Lobaplatin

INTERVENTIONS:
Drug: Lobaplatin — Patients enrolled will receive lobaplatin 30mg/m2 d1+ 5-FU 0.5g/m2/d d2-5 in every 21days. 4-6 cycles of chemotherapy are recommended.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of chemotherapy with Lobaplatin and 5-FU, in Recurrent Local or Distant Advanced Nasopharyngeal Carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* NPC diagnosed by pathology, with measurable lesions and imaging results, such as MRI and CT. Patients with no other lesions but bone metastasis are excluded.
* Recurrent locally or distant advanced NPC (rT3-4N0-3M0-1)
* ECOG 0 or 1
* Expected survival ≥ 1 year
* Without dysfunction of heart, lung, liver, kidney and hematopoiesis
* Patients are voluntary and signed informed consent
* No other anti-tumor treatment (including steroid)

Exclusion Criteria:

* Allergy history to platinum
* Use of 5-FU in last 6 months
* Had major surgery in last 4 weeks, or the wound has not completely healed
* Toxicity from previous treatment is still ≥CTC AE grade 3
* History of other carcinoma in the past 5 years, except for treated carcinoma in situ of cervix, as well as basal cell carcinoma or squamous cell carcinoma of the skin
* Dysfunction of heart
* Bleeding ≥CTC AE grade 3
* Use of anticoagulant or vitamin K antagonists, except for small dose of aspirin and warfarin for prevention
* Patients participated in clinical trials of other drugs within last 4 weeks
* Mental illness

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-07 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 2 years after chemotherapy
  the time from randomization to death or disease progression

SECONDARY OUTCOMES:
overall survival | 2 years after chemotherapy
  the time from randomization to death of any cause
objective response rate | 2 years after chemotherapy
  the ratio that patients who get PR or CR in all the patients

CONTACTS AND LOCATIONS:
Overall Officials: Yun-fei Xia, Professor, Principal Investigator — Department of Radiation Oncology, Sun Yat-Sen University Cancer Center
Locations (1):
- Department of Radiation Oncology, Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China